CLINICAL TRIAL: NCT03087149
Title: Supplementation of Vitamin D in Preterm Infants- Monitored Therapy vs Standard Therapy. A Randomized Controlled Trial
Brief Title: Monitored vs Standard Supplementation of Vitamin D in Preterm Infants
Acronym: MOSVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Anna Mazowiecka Hospital, Warsaw, Poland (Other)
Collaborators: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Alicja Kołodziejczyk, PhD student, Princess Anna Mazowiecka Hospital, Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VitD-2016
Record Dates: First submitted 2017-03-15; First posted 2017-03-22 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Vitamin D Deficiency; Osteopenia; Nephrolithiasis; Drug Overdose
Keywords: vitamin D; supplementation; hydroxyvitamin D; pretrem infants; osteopenia
MeSH Terms: conditions — Vitamin D Deficiency; Bone Diseases, Metabolic; Nephrolithiasis; Drug Overdose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- monitored group (Experimental): The monitored group will received monitored vit D supplementation
  Interventions: Dietary Supplement: monitored vit D supplementation
- standard group (Active Comparator): The standard group will receive standard vit D supplementation
  Interventions: Dietary Supplement: standard vit D supplementation

INTERVENTIONS:
Dietary Supplement: monitored vit D supplementation — The vit D supplementation dose start from dose 500IU from 7th day of age and is modified based on vit D measurement at 4 week of age for infants born <30 GA, at 8 week of age for infants born <26 GA at 35+/-2 weeks PMA(postmenstrual age), +/-at 40+/-2 weeks PMA according to the protocol.
  Arms: monitored group
Dietary Supplement: standard vit D supplementation — The vitamin D supplementation dose is 500IU from 7th day of age.
  Arms: standard group

SUMMARY:
The purpose of this study is to determine wheather the monitored vitamin D (vit D) therapy is safer and more effective than standard therapy in pretrem infants.

DETAILED DESCRIPTION:
Vitamin D (vit D) deficiency is a risk factor of osteopenia of prematurity, which leads to rickets or decreased bone mass mineral density. Recently multiple studies have been published on vit D adjust biological functions. Dosage, safety and effectiveness of vitD supplementation in preterm infants still remains a controversial topic. We hypothesize that monitored supplementation of vit D is more effective and safer than standard therapy 500IU in preterm infants. The study will be carried out in 138 preterm infants, born at 24-32 week of gestational age (GA) at the Princess Anne's Hospital in Warsaw, Poland. We will determine if monitored supplementation of vit D decreases the incidence of vit D deficiency and/or overdosing at 40 week (GA). For secondary objective we shall assess if monitored therapy reduces the incidence of vit D deficiency and/or overdosing at 35, 52 week (GA), prevalence of osteopenia, low bone mass, nephrocalcinosis and nephrolithiasis.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born between 24 and 32 weeks of gestation (estimated by ultrasound)
* In born or admitted to the unit within 48hours from birth.
* Randomization within 7 days from birth.
* Parental consent.
* Mothers willing to return for follow up visits.

Exclusion Criteria:

* Preterm delivery >=33 weeks of gestation or term delivery (estimated by ultrasound).
* Major congenital abnormalities.
* Participation in another trial.
* Severe illness at birth deemed incompatible with survival.
* Congenital HIV infection.
* Total parenteral nutrition > 14 days.
* Cholestasis

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with D- deficiency or access | at 40 (+/-2 weeks) PMA (postmenstrual age)
  25-hydroxyvitamin D serum level below 20ng/ml (50nmol/l ) or above 100ng/ml (250nmol/l )
Number of Participants with D- deficiency or access | at 4 weeks of age
  25-hydroxyvitamin D serum level below 20ng/ml (50nmol/l ) or above 100ng/ml (250nmol/l )
Number of Participants with D- deficiency or access | At 35 (+/-2 weeks) PMA (postmenstrual age)
  25-hydroxyvitamin D serum level below 20ng/ml (50nmol/l ) or above 100ng/ml (250nmol/l )
Number of Participants with D- deficiency or access | At 52 (+/-2 weeks) PMA (postmenstrual age)
  25-hydroxyvitamin D serum level below 20ng/ml (50nmol/l ) or above 100ng/ml (250nmol/l )

SECONDARY OUTCOMES:
Number of Participants with biochemical markers of osteopenia | at 35, 40, 52 (+/-2 weeks) PMA (postmenstrual age)
  ALP>500IU and serum phosphate level <1,8mmol/l or ALP>900IU
average of bone mass | at 35, 40 (+/-2 weeks) PMA
  measurement of speed of sound [SOS] in meters per second in the axial transmission mode with a small ultrasound probe along the mid tibia by Sunlight Omnisence 7000 Premier using CRB Probe
Number of Participants with hypercalcemia | at 35, 40, 52 (+/-2 weeks) PMA (postmenstrual age)
  serum calcium level above 2,75mmol/l
Number of Participants with hypercalcuria | at 35, 40, 52 (+/-2 weeks) PMA
  urine calcium:creatinine ratio >3,8mmol/mmol for 0-4 week of age; >3,5mmol/mmol for 5-8 week of age; >2,8mmol/mmol for 9-12 week of age; >2,5mmol/mmol for 13-18 week of age; >2,2mmol/mmol for >19 week of age
Number of Participants with nephrocalcinosis | at 35, 52 (+/-2 weeks) PMA
  nephrocalcinosis detected in ultrasonography examination of kidneys

OTHER OUTCOMES:
Number of Participants with vitamin D- acceptable range | at 35, 40, 52 (+/-2 weeks) PMA (postmenstrual age)
  25-hydroxyvitamin D serum level between 30ng/ml (75nmol/l ) and 80ng/ml (200nmol/l )
Number of Participants with vitamin D- optimal range | at 35, 40, 52 (+/-2 weeks) PMA (postmenstrual age)
  25-hydroxyvitamin D serum level between 30ng/ml (75nmol/l ) and 50ng/ml (125nmol/l )
Avarage of vitamin D level | at 35, 40, 52 (+/-2 weeks) PMA (postmenstrual age)
  25-hydroxyvitamin D serum level

CONTACTS AND LOCATIONS:
Overall Officials: Maria K Borszewska-Kornacka, Professor, Study Chair — Princess Anna Mazowiecka Hospital; Renata Bokiniec, M.D., Study Director — Princess Anna Mazowiecka Hospital
Locations (1):
- Princess Anna Mazowiecka Hospital, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Backstrom MC, Maki R, Kuusela AL, Sievanen H, Koivisto AM, Ikonen RS, Kouri T, Maki M. Randomised controlled trial of vitamin D supplementation on bone density and biochemical indices in preterm infants. Arch Dis Child Fetal Neonatal Ed. 1999 May;80(3):F161-6. doi: 10.1136/fn.80.3.f161. PMID 10212074
- [Background] Rigo J, Pieltain C, Salle B, Senterre J. Enteral calcium, phosphate and vitamin D requirements and bone mineralization in preterm infants. Acta Paediatr. 2007 Jul;96(7):969-74. doi: 10.1111/j.1651-2227.2007.00336.x. PMID 17577338
- [Background] Zerofsky M, Ryder M, Bhatia S, Stephensen CB, King J, Fung EB. Effects of early vitamin D deficiency rickets on bone and dental health, growth and immunity. Matern Child Nutr. 2016 Oct;12(4):898-907. doi: 10.1111/mcn.12187. Epub 2015 Apr 7. PMID 25850574
- [Background] Zhu K, Whitehouse AJ, Hart PH, Kusel M, Mountain J, Lye S, Pennell C, Walsh JP. Maternal vitamin D status during pregnancy and bone mass in offspring at 20 years of age: a prospective cohort study. J Bone Miner Res. 2014;29(5):1088-95. doi: 10.1002/jbmr.2138. PMID 24189972
- [Background] Dinlen N, Zenciroglu A, Beken S, Dursun A, Dilli D, Okumus N. Association of vitamin D deficiency with acute lower respiratory tract infections in newborns. J Matern Fetal Neonatal Med. 2016 Mar;29(6):928-32. doi: 10.3109/14767058.2015.1023710. Epub 2015 Mar 19. PMID 25786473
- [Background] Grant CC, Kaur S, Waymouth E, Mitchell EA, Scragg R, Ekeroma A, Stewart A, Crane J, Trenholme A, Camargo CA Jr. Reduced primary care respiratory infection visits following pregnancy and infancy vitamin D supplementation: a randomised controlled trial. Acta Paediatr. 2015 Apr;104(4):396-404. doi: 10.1111/apa.12819. Epub 2014 Oct 21. PMID 25283480
- [Background] Gernand AD, Simhan HN, Caritis S, Bodnar LM. Maternal vitamin D status and small-for-gestational-age offspring in women at high risk for preeclampsia. Obstet Gynecol. 2014 Jan;123(1):40-48. doi: 10.1097/AOG.0000000000000049. PMID 24463662
- [Background] Whitehouse AJ, Holt BJ, Serralha M, Holt PG, Kusel MM, Hart PH. Maternal serum vitamin D levels during pregnancy and offspring neurocognitive development. Pediatrics. 2012 Mar;129(3):485-93. doi: 10.1542/peds.2011-2644. Epub 2012 Feb 13. PMID 22331333
- [Background] Pludowski P, Holick MF, Pilz S, Wagner CL, Hollis BW, Grant WB, Shoenfeld Y, Lerchbaum E, Llewellyn DJ, Kienreich K, Soni M. Vitamin D effects on musculoskeletal health, immunity, autoimmunity, cardiovascular disease, cancer, fertility, pregnancy, dementia and mortality-a review of recent evidence. Autoimmun Rev. 2013 Aug;12(10):976-89. doi: 10.1016/j.autrev.2013.02.004. Epub 2013 Mar 28. PMID 23542507
- [Background] Vogiatzi MG, Jacobson-Dickman E, DeBoer MD; Drugs, and Therapeutics Committee of The Pediatric Endocrine Society. Vitamin D supplementation and risk of toxicity in pediatrics: a review of current literature. J Clin Endocrinol Metab. 2014 Apr;99(4):1132-41. doi: 10.1210/jc.2013-3655. Epub 2014 Jan 23. PMID 24456284
- [Background] Javaid MK, Crozier SR, Harvey NC, Gale CR, Dennison EM, Boucher BJ, Arden NK, Godfrey KM, Cooper C; Princess Anne Hospital Study Group. Maternal vitamin D status during pregnancy and childhood bone mass at age 9 years: a longitudinal study. Lancet. 2006 Jan 7;367(9504):36-43. doi: 10.1016/S0140-6736(06)67922-1. PMID 16399151
- [Background] Hollis BW, Johnson D, Hulsey TC, Ebeling M, Wagner CL. Vitamin D supplementation during pregnancy: double-blind, randomized clinical trial of safety and effectiveness. J Bone Miner Res. 2011 Oct;26(10):2341-57. doi: 10.1002/jbmr.463. Erratum In: J Bone Miner Res. 2011 Dec; 26(12):3001. PMID 21706518
- [Background] Whitehouse AJ, Holt BJ, Serralha M, Holt PG, Hart PH, Kusel MM. Maternal vitamin D levels and the autism phenotype among offspring. J Autism Dev Disord. 2013 Jul;43(7):1495-504. doi: 10.1007/s10803-012-1676-8. PMID 23070790
- [Background] Cetinkaya M, Cekmez F, Erener-Ercan T, Buyukkale G, Demirhan A, Aydemir G, Aydin FN. Maternal/neonatal vitamin D deficiency: a risk factor for bronchopulmonary dysplasia in preterms? J Perinatol. 2015 Oct;35(10):813-7. doi: 10.1038/jp.2015.88. Epub 2015 Jul 30. PMID 26226242
- [Background] Cizmeci MN, Kanburoglu MK, Akelma AZ, Ayyildiz A, Kutukoglu I, Malli DD, Tatli MM. Cord-blood 25-hydroxyvitamin D levels and risk of early-onset neonatal sepsis: a case-control study from a tertiary care center in Turkey. Eur J Pediatr. 2015 Jun;174(6):809-15. doi: 10.1007/s00431-014-2469-1. Epub 2014 Dec 12. PMID 25504199
- [Background] Abrams SA; Committee on Nutrition. Calcium and vitamin d requirements of enterally fed preterm infants. Pediatrics. 2013 May;131(5):e1676-83. doi: 10.1542/peds.2013-0420. Epub 2013 Apr 29. PMID 23629620
- [Background] Agostoni C, Buonocore G, Carnielli VP, De Curtis M, Darmaun D, Decsi T, Domellof M, Embleton ND, Fusch C, Genzel-Boroviczeny O, Goulet O, Kalhan SC, Kolacek S, Koletzko B, Lapillonne A, Mihatsch W, Moreno L, Neu J, Poindexter B, Puntis J, Putet G, Rigo J, Riskin A, Salle B, Sauer P, Shamir R, Szajewska H, Thureen P, Turck D, van Goudoever JB, Ziegler EE; ESPGHAN Committee on Nutrition. Enteral nutrient supply for preterm infants: commentary from the European Society of Paediatric Gastroenterology, Hepatology and Nutrition Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2010 Jan;50(1):85-91. doi: 10.1097/MPG.0b013e3181adaee0. PMID 19881390
- [Background] Pludowski P, Karczmarewicz E, Bayer M, Carter G, Chlebna-Sokol D, Czech-Kowalska J, Debski R, Decsi T, Dobrzanska A, Franek E, Gluszko P, Grant WB, Holick MF, Yankovskaya L, Konstantynowicz J, Ksiazyk JB, Ksiezopolska-Orlowska K, Lewinski A, Litwin M, Lohner S, Lorenc RS, Lukaszkiewicz J, Marcinowska-Suchowierska E, Milewicz A, Misiorowski W, Nowicki M, Povoroznyuk V, Rozentryt P, Rudenka E, Shoenfeld Y, Socha P, Solnica B, Szalecki M, Talalaj M, Varbiro S, Zmijewski MA. Practical guidelines for the supplementation of vitamin D and the treatment of deficits in Central Europe - recommended vitamin D intakes in the general population and groups at risk of vitamin D deficiency. Endokrynol Pol. 2013;64(4):319-27. doi: 10.5603/ep.2013.0012. PMID 24002961
- [Background] Monangi N, Slaughter JL, Dawodu A, Smith C, Akinbi HT. Vitamin D status of early preterm infants and the effects of vitamin D intake during hospital stay. Arch Dis Child Fetal Neonatal Ed. 2014 Mar;99(2):F166-8. doi: 10.1136/archdischild-2013-303999. Epub 2013 Jul 13. PMID 23852093
- [Background] Pinto K, Collins CT, Gibson RA, Andersen CC. Vitamin D in preterm infants: A prospective observational study. J Paediatr Child Health. 2015 Jul;51(7):679-81. doi: 10.1111/jpc.12847. Epub 2015 Feb 12. PMID 25683497
- [Background] Fort P, Salas AA, Nicola T, Craig CM, Carlo WA, Ambalavanan N. A Comparison of 3 Vitamin D Dosing Regimens in Extremely Preterm Infants: A Randomized Controlled Trial. J Pediatr. 2016 Jul;174:132-138.e1. doi: 10.1016/j.jpeds.2016.03.028. Epub 2016 Apr 11. PMID 27079965
- [Background] Backstrom MC, Kouri T, Kuusela AL, Sievanen H, Koivisto AM, Ikonen RS, Maki M. Bone isoenzyme of serum alkaline phosphatase and serum inorganic phosphate in metabolic bone disease of prematurity. Acta Paediatr. 2000 Jul;89(7):867-73. PMID 10943972
- [Background] Nemet D, Dolfin T, Wolach B, Eliakim A. Quantitative ultrasound measurements of bone speed of sound in premature infants. Eur J Pediatr. 2001 Dec;160(12):736-40. doi: 10.1007/s004310100849. PMID 11795683
- [Background] Rack B, Lochmuller EM, Janni W, Lipowsky G, Engelsberger I, Friese K, Kuster H. Ultrasound for the assessment of bone quality in preterm and term infants. J Perinatol. 2012 Mar;32(3):218-26. doi: 10.1038/jp.2011.82. Epub 2011 Jun 16. PMID 21681177
- [Derived] Kolodziejczyk A, Borszewska-Kornacka MK, Seliga-Siwecka J. MOnitored supplementation of VItamin D in preterm infants (MOSVID trial): study protocol for a randomised controlled trial. Trials. 2017 Sep 11;18(1):424. doi: 10.1186/s13063-017-2141-y. PMID 28893306
- See also: Related Info — http://www.yeec.com/uploadimages1/forum/kone/konelabreferencemanual.pdf